CLINICAL TRIAL: NCT04629183
Title: Risk Stratification of COVID-19 Patients Discharged From the Emergency Department
Acronym: CODED
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Fulvio Morello, Associate Professor (Internal Medicine), S.C. Medicina d'Urgenza U (MECAU), Università degli Studi di Torino, A.O.U. Città della Salute e della Scienza
Other Study IDs: COVID-ED-IntRisk
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: emergency department; admission; discharge; risk
MeSH Terms: conditions — COVID-19; Emergencies | interventions — X-Rays; Standard of Care; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: integrated clinical evaluation — 30-day follow-up (telephone/database query) to define outcome Patients will receive standard care, independent of study participation.
  Other Names: lung ultrasonosgraphy; chest radiography (standard care, clinical decision); blood testing (standard care, clinical decision)

SUMMARY:
Risk stratification of COVID-19 patients is essential to define their appropriate treatment setting. So far, available studies have focused on morbidity and mortality prediction in patients admitted to hospital. In the Emergency Department (ED), decision on home discharge versus hospital admission for COVID-19 is cumbersome. While facing a dramatic second wave of SARS-CoV-2, shortage of hospital beds has further increased the challenge.

The present study will prospectively evaluate the clinical outcomes of patients discharged from the ED. Stratification will be based on a composite of demographic, clinical and lung imaging variables. Results will be used to develop standardized decision rules for safe home discharge of patients with COVID-19 evaluated in the ED.

DETAILED DESCRIPTION:
Patients with inclusion criteria and without exclusion criteria, evaluated in the participating EDs, will be enrolled in the study. Patients will undergo standard medical evaluation by the attending physician(s), following local guidelines and best medical practice, independent of participation to the study.

The following data will be recorded, when available:

* Demographic/clinical: age, gender, symptoms (type, time from onset), comorbidities, Glasgow Coma Scale score, respiratory rate, peripheral oxygen saturation
* Biochemical: urea, creatinine, C-reactive protein, procalcitonin, lactate dehydrogenase, white blood cell count, lymphocyte count, d-dimer
* Lung ultrasonography: site/type of B lines, consolidations, pleural effusion
* Radiology: chest X-ray result, chest CT result

Upon discharge, patients will be encouraged to contact emergency medical services or return the ED if needed, in case of clinical worsening.

The following endpoint will be assessed at 30 days after ED discharge, through standardized telephone interview and healthcare/other database query: any further hospital admission (for COVID-19 or other disease), death (for COVID-19 or other disease), respiratory failure/ventilation/intensive care admission (only for hospitalized COVID-19 patients).

Data analysis will focus on the outcome incidence in the study cohort, stratified by a composite of demographic/clinical, biochemical and imaging variables. A key stratification tool will be the 4C mortality score (BMJ 2020; 370 doi: https://doi.org/10.1136/bmj.m3339). Additional integration of study variables will be evaluated to improve stratification and prediction.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic COVID-19 confirmed by treating physician
* positive nasopharyngeal swab for SARS-CoV-2 (performed during the ED visit or within last 14 days)
* First ED visit for suspected or confirmed COVID-19 (within last 30 days)
* Home discharge from ED based on treating physician's or patient's decision

Exclusion Criteria:

* Age <18 years
* Nursing home resident
* Already on home oxygen therapy
* Previous ED visit for suspected or confirmed COVID-19 (within last 30 days)
* Informed consent denial
* Follow-up not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years) subjected to a first ED visit for physician-confirmed COVID-19, discharged from the ED based on attending physician's or patient's decision (independent from study participation). Patients will provide their informed consent to participation (thus allowing clinical data recording and 30-day follow-up).
Sampling Method: Non-Probability Sample
Enrollment: 742 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
composite outcome | 30 days
  death (any cause), hospital admission (any cause)

SECONDARY OUTCOMES:
death (COVID-19) | 30 days
  death for COVID-19
death (other disease) | 30 days
  death for disease other than COVID-19
hospital admission (COVID-19) | 30 days
  subsequent hospital admission for COVID-19
hospital admission (other disease) | 30 days
  subsequent hospital admission for disease other than COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Morello, MD, PhD, Principal Investigator — A.O.U. Città della Salute e della Scienza di Torino
Locations (7):
- Italy (7):
  - Ospedale Maria Vittoria, D.E.A., Turin, Piedmont
  - A.O.U.C. Azienda Ospedaliero-Universitaria Careggi, D.E.A., Florence, Tuscany
  - Ospedale U. Parini, Medicina e Chirurgia d'accettazione e Urgenza (MeCAU), Aosta
  - A.O. S. Croce e Carle, Medicina e Chirurgia d'Urgenza, Cuneo
  - A.O.U. Careggi, Medicina e Chirurgia d'Urgenza e Accettazione, Florence
  - A.O.U. Città della Salute e della Scienza di Torino, Ospedale Molinette, S.C. Medicina d'Urgenza U (MECAU), Torino
  - Ospedale San Giovanni Bosco, Medicina e Chirurgia d'accettazione e urgenza (MeCAU), Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pivetta E, Goffi A, Tizzani M, Locatelli SM, Porrino G, Losano I, Leone D, Calzolari G, Vesan M, Steri F, Arianna A, Capuano M, Gelardi M, Silvestri G, Dutto S, Avolio M, Cavallo R, Bartalucci A, Paglieri C, Morello F, Richiardi L, Maule MM, Lupia E, on behalf of the Molinette MedUrg Group on Lung Ultrasound. Lung ultrasound for the diagnosis of SARS-CoV-2 pneumonia in the Emergency Department. https://doi.org/10.1016/j.annemergmed.2020.10.008
- [Result] Knight SR, Ho A, Pius R, Buchan I, Carson G, Drake TM, Dunning J, Fairfield CJ, Gamble C, Green CA, Gupta R, Halpin S, Hardwick HE, Holden KA, Horby PW, Jackson C, Mclean KA, Merson L, Nguyen-Van-Tam JS, Norman L, Noursadeghi M, Olliaro PL, Pritchard MG, Russell CD, Shaw CA, Sheikh A, Solomon T, Sudlow C, Swann OV, Turtle LC, Openshaw PJ, Baillie JK, Semple MG, Docherty AB, Harrison EM; ISARIC4C investigators. Risk stratification of patients admitted to hospital with covid-19 using the ISARIC WHO Clinical Characterisation Protocol: development and validation of the 4C Mortality Score. BMJ. 2020 Sep 9;370:m3339. doi: 10.1136/bmj.m3339. PMID 32907855
- [Result] Liu RB, Tayal VS, Panebianco NL, Tung-Chen Y, Nagdev A, Shah S, Pivetta E, Henwood PC, Nelson MJ, Moore CL. Ultrasound on the Frontlines of COVID-19: Report From an International Webinar. Acad Emerg Med. 2020 Jun;27(6):523-526. doi: 10.1111/acem.14004. Epub 2020 Jun 9. No abstract available. PMID 32348585